CLINICAL TRIAL: NCT01857323
Title: A Prospective, Open-Label Assessment of the Albuterol Spiromax® DPI Integrated Dose Counter
Brief Title: Open-Label Assessment of the Albuterol Spiromax® Dry Powder Inhaler (DPI)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ABS-AS-308
Record Dates: First submitted 2013-05-15; First posted 2013-05-20 (Estimated); Results first posted 2015-06-08 (Estimated); Last update posted 2015-06-08 (Estimated); Status verified 2015-05

CONDITIONS: Asthma; Chronic Obstructive Pulmonary Disease (COPD)
Keywords: asthma; chronic obstructive pulmonary disease; COPD; Albuterol Spiromax®
MeSH Terms: conditions — Asthma; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Albuterol Spiromax® (Experimental): The approximate 50-day treatment period consisted of 180 mcg (90 mcg/dose cycle, 2 dose cycles) twice daily study medication administration with Albuterol Spiromax with dose-counter.
  Interventions: Drug: Albuterol Spiromax®

INTERVENTIONS:
Drug: Albuterol Spiromax® — Albuterol Spiromax delivers 90 mcg of albuterol base from the mouthpiece per triggered dose. Participants took doses of 2 inhalations each twice a day (morning and evening) for a total daily dose of 360 mcg. The first 45 enrolled participants constituted a subgroup who were dosed for 35 days, while most participants were dosed for 50 days.
  Other Names: ProAir® RespiClick, Albuterol multi-dose dry powder inhaler (MDPI)

SUMMARY:
This is a prospective, open-label, multicenter Phase 3 study evaluating the performance of the Albuterol Spiromax dose counter in patients with a diagnosis of asthma and/or COPD. The purpose of this study is to evaluate the functionality, reliability, and accuracy of the Albuterol Spiromax inhaler integrated dose counter in a clinical setting.

DETAILED DESCRIPTION:
The study consists of a screening/run-in period where, after meeting study criteria, patients enter a run-in period lasting 7 to 14 ±2 days, during which diary and medication compliance, as well as inhaler technique, will be assessed. The run-in period will commence the day following the completion of all screening procedures and will continue through to and include the day prior to the first treatment visit (TV1) such that a minimum of 7 full days of diary data will be collected prior to TV1. The purpose of the run-in period is to assess compliance with a BID dosing regimen and with the completion of the diary entries over a minimum period of 7 days. Patients who demonstrate adequate inhaler technique and who are at least 90% compliant with dosing and completion of the diary on the last 7 consecutive days of run-in will qualify for enrollment into the open-label study. The study treatment period will comprise 6 treatment visits (TV1-TV6) for all enrolled patients except those in the 5-week treatment cohort who will have only 5 treatment visits (TV1-TV5). Patients may continue taking their current asthma or COPD medications throughout the Treatment Period. The patient will return to the clinic on Days 8 (±1), 15 (±1), 22 (±1), and 36 (±1), and then on Day 50 (-2) after approximately all 200 doses have been delivered, or until early withdrawal. The patient will be deemed to have completed the study if at least 90% of the recommended doses contained in Albuterol Spiromax with dose-counter were used. A representative sample (approximately 15%) of patients will participate in the trial for approximately 5 weeks with Day 36 (±1) being the final study visit.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent/assent signed and dated by the patient and/or parent/legal guardian before conducting any study related procedure
2. Male or female (non pregnant/non lactating) patients 4 years of age or older at the time of the screening visit (SV) who are able to understand English
3. Females of childbearing potential (as judged by the investigator) currently using and will continue to use a medically reliable method of contraception for the entire study duration (e.g. oral, injectable, trans-cutaneous or implantable contraceptives or intrauterine devices or double-barrier protection). Females who are not sexually active must agree to use a medically reliable method of contraception should they become active during the course of the study. Women of childbearing potential, or less than 1 year postmenopausal, will require a negative urine pregnancy test at the SV. Female patients will be considered to be of non-child-bearing potential and will not require a urine pregnancy test if at least one of the following apply:a. before menarche; b. more than one year post-menopausal; c. had a hysterectomy, bilateral oophorectomy, salpingectomy, or tubal ligation; d. has congenital sterility
4. General good health, defined as free of any concomitant conditions or treatment that could interfere with study conduct, influence the interpretation of study observations/results, or put the patient at increased risk during the study
5. Has a physician diagnosis of asthma or COPD with symptoms of bronchoconstriction requiring the use of short-acting β2-agonists
6. Current Therapy: The patient's current asthma/COPD controller treatment regimen has remained stable for at least four weeks prior to the SV
7. Capable of understanding the requirements, risks, and benefits of study participation, and, as judged by the investigator, capable of giving informed consent/assent and being compliant with all study requirements (visits, record keeping, etc)
8. Able to demonstrate satisfactory Spiromax inhaler use and technique.

Exclusion Criteria:

1. History of life-threatening asthma or COPD that is defined for this protocol as an asthma or COPD episode that required intubation and/or was associated with hypercapnea, respiratory arrest, or hypoxic seizures
2. Culture-documented or suspected bacterial or viral infection of the upper or lower respiratory tract, sinus, or middle ear that is not resolved within 2 weeks of the SV; or that occurs between the SV and TV1
3. Is being treated with a long-acting β2-agonist alone
4. Any asthma exacerbation requiring oral corticosteroids within 2 months of SV and any COPD exacerbation requiring oral corticosteroids within 1 month of the SV. A patient must not have been hospitalized for asthma or COPD within 4 months prior to the SV.
5. Historical or current evidence of a clinically significant disease including, but not limited to: cardiovascular (e.g., congestive heart failure, known aortic aneurysm, clinically significant cardiac arrhythmia or coronary heart disease, cerebrovascular accident), hepatic, renal, hematological, neuropsychological, endocrine (e.g., uncontrolled diabetes mellitus, uncontrolled thyroid disorder, Addison's disease, Cushing's syndrome), and/or gastrointestinal (e.g., poorly-controlled peptic ulcer or gastroesophageal reflux disease [GERD]). Significant is defined as any disease that, in the opinion of the investigator, would put the safety of the patient at risk through participation, or which could affect the endpoint analysis if the disease/condition exacerbated during the study.
6. Uncontrolled hypertension (systolic blood pressure [BP] ≥160 mmHg or diastolic BP >100 mmHg)
7. History of any adverse reaction, including immediate or delayed hypersensitivity to any β2-agonist, sympathomimetic drug, or any component of the Albuterol Spiromax DPI or rescue ProAir Hydrofluoroalkane (HFA) Metered-dose inhaler (MDI) formulation.
8. Other exclusion criteria apply.

Min Age: 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 317 (Actual)
Dates: Start 2013-05; Primary Completion 2013-08 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (30):
- United States (30):
  - Teva Investigational Site 10620, Phoenix, Arizona
  - Teva Investigational Site 10637, Costa Mesa, California
  - Teva Investigational Site 10635, Huntington Beach, California
  - Teva Investigational Site 10647, Rolling Hills Estates, California
  - Teva Investigational Site 10643, San Diego, California
  - Teva Investigational Site 10644, San Jose, California
  - Teva Investigational Site 10622, Centennial, Colorado
  - Teva Investigational Site 10634, Denver, Colorado
  - Teva Investigational Site 10645, Wheat Ridge, Colorado
  - Teva Investigational Site 10633, Miami, Florida
  - Teva Investigational Site 10640, Ormond Beach, Florida
  - Teva Investigational Site 10641, Overland Park, Kansas
  - Teva Investigational Site 10636, Bethesda, Maryland
  - Teva Investigational Site 10631, North Dartmouth, Massachusetts
  - Teva Investigational Site 10646, Plymouth, Minnesota
  - Teva Investigational Site 10627, St Louis, Missouri
  - Teva Investigational Site 10642, Bozeman, Montana
  - Teva Investigational Site 10613, High Point, North Carolina
  - Teva Investigational Site 10616, Raleigh, North Carolina
  - Teva Investigational Site 10618, Canton, Ohio
  - Teva Investigational Site 10615, Oklahoma City, Oklahoma
  - Teva Investigational Site 10624, Tulsa, Oklahoma
  - Teva Investigational Site 10625, Eugene, Oregon
  - Teva Investigational Site 10626, Medford, Oregon
  - Teva Investigational Site 10632, Portland, Oregon
  - Teva Investigational Site 10639, Charleston, South Carolina
  - Teva Investigational Site 10617, Spartanburg, South Carolina
  - Teva Investigational Site 10630, Dallas, Texas
  - Teva Investigational Site 10623, New Braunfels, Texas
  - Teva Investigational Site 10638, San Antonio, Texas

REFERENCES:
- [Derived] Given J, Taveras H, Iverson H. Prospective, open-label evaluation of a new albuterol multidose dry powder inhaler with integrated dose counter. Allergy Asthma Proc. 2016 May;37(3):199-206. doi: 10.2500/aap.2016.37.3938. Epub 2016 Jan 29. PMID 26831652

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of the 28 screened patients who were not enrolled, 12 were excluded on the basis of inclusion criteria, 7 patients for exclusion criteria, 4 patients withdrew consent,1 patient was non-compliant, and 4 patients withdrew for other reasons before the baseline visit.
Period: Overall Study
Arm/Group | Albuterol Spiromax®
Started | 317 (36 day treatment cohort: 45 participants 50 day treatment cohort: 272 participants)
Safety Population | 316 (One enrolled participant was lost to follow-up.)
Completed | 253
Not Completed | 64
Not completed — Adverse Event | 1
Not completed — Withdrawal by Subject | 3
Not completed — Non-compliance | 1
Not completed — Protocol Violation | 6
Not completed — Lost to Follow-up | 1
Not completed — Other | 4
Not completed — Did not complete 180 doses | 48

BASELINE CHARACTERISTICS:
Population: ITT population
Arm/Group | Albuterol Spiromax®
Number analyzed (Participants) | 317
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.3 (22.7)
Age, Customized [Number; unit: participants]
  4-11 years | 44
  12-64 years | 144
  65+ years | 129
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 178
  Male | 139
Race/Ethnicity, Customized [Number; unit: participants]
  White | 268
  Black | 35
  Asian | 7
  American Indian or Alaskan Native | 1
  Pacific Islander | 1
  Other, not specified | 5
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic or Latino | 25
  Non-Hispanic, non-Latino | 292
Disease Type [Number; unit: participants] — COPD = Chronic obstructive pulmonary disease
  participants
    Asthma | 167
    COPD | 150

OUTCOME MEASURES:

1. Primary Outcome: Dosing Discrepancies Per 200 Dose Cycles: Dose Cycle Not Count
Description: The purpose of the study is to determine if the dose counter on Albuterol Spiromax is counting accurately; accuracy is determined by concordance/agreement between patient-reported Albuterol Spiromax counter readings and patient-reported dose cycles recorded in patient diaries. This outcome measures how often the dose cycle was not counted: the participant completes a full dose cycle (opens the mouthpiece cap, inhales the medication, and closes the mouthpiece cap) but the counter display does not advance (i.e., does not count down) within a dosing session. The discrepancy rate was calculated as "number of discrepancies/total number of dose cycles" *200.
Time Frame: Day 1 - Day 50
Population: Per protocol population includes all data from randomized participants who have not experienced major protocol violations prior to dosing with at least 180 inhaled doses. Participants in the 35-day subgroup are excluded from the PP population, as they will only have taken approximately 140 doses during the study.
Measure: Number; unit: discrepancies/200 dose cycles
Units Other Than Participants: Total # of dose cycles
Arm/Group | Albuterol Spiromax®
Number analyzed (Participants) | 253
Number analyzed (Total # of dose cycles) | 49454
discrepancies/200 dose cycles | 2.05

2. Secondary Outcome: Dosing Discrepancies Per 200 Dose Cycles: Dose Cycle Count Up
Description: The purpose of the study is to determine if the dose counter on Albuterol Spiromax is counting accurately; accuracy is determined by concordance/agreement between patient-reported Albuterol Spiromax counter readings and patient-reported dose cycles recorded in patient diaries. This outcome measures when the inhaler counter reading increases, instead of decreases, after the participant has executed the dose cycle (i.e., the ending counter reading is greater than the beginning counter reading within a dosing session). The discrepancy rate was calculated as "number of discrepancies/total number of dose cycles" *200.
Time Frame: Day 1 - Day 50
Population: as for outcome 1
Measure: Number; unit: discrepancies/200 dose cycles
Units Other Than Participants: Total # of dose cycles
Arm/Group | Albuterol Spiromax®
Number analyzed (Participants) | 253
Number analyzed (Total # of dose cycles) | 49454
discrepancies/200 dose cycles | 2.46

3. Secondary Outcome: Dosing Discrepancies Per 200 Dose Cycles: Count Unknown Dose Cycle
Description: The purpose of the study is to determine if the dose counter on Albuterol Spiromax is counting accurately; accuracy is determined by concordance/agreement between patient-reported Albuterol Spiromax counter readings and patient-reported dose cycles recorded in patient diaries. This outcome measures when the inhaler counter advances (decreases, e.g., 50 to 48) between dosing sessions but the participant has not knowingly executed the dose cycle (i.e., the counter number at the beginning of the dosing session is less than the counter number at the end of the previous dosing session). The discrepancy rate was calculated as "number of discrepancies/total number of dose cycles" *200.
Time Frame: Day 1 - Day 50
Population: as for outcome 1
Measure: Number; unit: discrepancies/200 dose cycles
Units Other Than Participants: Total # of dose cycles
Arm/Group | Albuterol Spiromax®
Number analyzed (Participants) | 253
Number analyzed (Total # of dose cycles) | 49454
discrepancies/200 dose cycles | 0.43

4. Secondary Outcome: Dosing Discrepancies Per 200 Dose Cycles: Count Up Unknown Dose Cycle
Description: The purpose of the study is to determine if the dose counter on Albuterol Spiromax is counting accurately; accuracy is determined by concordance/agreement between patient-reported Albuterol Spiromax counter readings and patient-reported dose cycles recorded in patient diaries. This outcome measures when the inhaler counter counts upwards (number increases, e.g. 50 to 52) rather than downward between dosing sessions but the participant has not knowingly executed the dose cycle (i.e., the counter number at the beginning of the dosing session is greater than the counter number at the end of the previous dosing session). The discrepancy rate was calculated as "number of discrepancies/total number of dose cycles" *200.
Time Frame: Day 1 - Day 50
Population: as for outcome 1
Measure: Number; unit: discrepancies/200 dose cycles
Units Other Than Participants: Total # of dose cycles
Arm/Group | Albuterol Spiromax®
Number analyzed (Participants) | 253
Number analyzed (Total # of dose cycles) | 49454
discrepancies/200 dose cycles | 0.17

5. Secondary Outcome: Absolute Value of Total Discrepancy Size Per Inhaler
Description: The purpose of the study is to determine if the dose counter on Albuterol Spiromax is counting accurately; accuracy is determined by concordance/agreement between patient-reported Albuterol Spiromax counter readings and patient-reported dose cycles recorded in patient diaries. This outcome is calculated for each inhaler as "beginning counter reading minus end counter reading" minus "patient-recorded number of dose cycles". The total inhaler discrepancy size is an important measure because it provides the most relevant means of ensuring that the inhaler does not exhaust its supply of albuterol before the counter has recorded the labeled 200 doses.
Time Frame: Day 1 - Day 50
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: discrepancies/inhaler
Arm/Group | Albuterol Spiromax®
Number analyzed (Participants) | 253
discrepancies/inhaler | 2.0 (2.88)

6. Secondary Outcome: Participants With Treatment-Emergent Adverse Events
Description: Adverse events (AEs) summarized in this table are those that began or worsened after treatment with study drug (treatment-emergent AEs). An adverse event was defined in the protocol as any untoward medical occurrence that develops or worsens in severity during the conduct of a clinical study and does not necessarily have a causal relationship to the study drug. Severity was rated by the investigator on a scale of mild, moderate and severe, with severe= an AE which prevents normal daily activities. Relation of AE to treatment was determined by the investigator. Serious AEs include death, a life-threatening adverse event, inpatient hospitalization or prolongation of existing hospitalization, persistent or significant disability or incapacity, a congenital anomaly or birth defect, OR an important medical event that jeopardized the patient and required medical intervention to prevent the previously listed serious outcomes.
Time Frame: Day 1 to Day 50
Population: Safety population
Measure: Number; unit: participants
Arm/Group | Albuterol Spiromax®
Number analyzed (Participants) | 316
participants
  Any adverse event | 85
  Severe adverse event | 2
  Treatment-related adverse event | 7
  Deaths | 0
  Other serious adverse events | 2
  Withdrawn from study due to adverse event | 1

ADVERSE EVENTS:
Time Frame: Day 1 to Day 50
Arm/Group | Albuterol Spiromax®
Serious Adverse Events (participants affected / at risk) | 2/316
Other Adverse Events (participants affected / at risk) | 15/316
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Albuterol Spiromax® (N=316)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 1 (1)
Drug eruption (Skin and subcutaneous tissue disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Albuterol Spiromax® (N=316)
Sinusitis (Infections and infestations) | 7 (7)
Headache (Nervous system disorders) | 8 (10)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor has the right 60 days before submission for publication to review/provide comments. If the Sponsor's review shows that potentially patentable subject matter would be disclosed, publication or public disclosure shall be delayed for up to 90 additional days in order for the Sponsor, or Sponsor's designees, to file the necessary patent applications. In multicenter trials, each PI will postpone single center publications until after disclosure or publication of multicenter data.